CLINICAL TRIAL: NCT03420716
Title: Effect of Regular Consumption of a Symbiotic Yogurt on Calcium Absorption and Bone Health in Young Adult Women
Brief Title: Symbiotic Yogurt, Calcium Absorption and Bone Health in Young Adult Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de la Republica (Other)
Responsible Party: Principal Investigator, Carmen Marino Donangelo, Professor, Universidad de la Republica
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: URepublica 01
Record Dates: First submitted 2018-01-12; First posted 2018-02-05 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Osteoporosis
Keywords: functional foods; dairy foods; calcium absorption; prebiotics and probiotics; young women; bone health
MeSH Terms: conditions — Osteoporosis | interventions — Yogurt

STUDY DESIGN:
Intervention Model Description: 3 weeks on symbiotic yogurt or control yogurt, with a 3 week wash out period in between. Type of yougurt consumed first is randomized.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Type of yogurt fed is blind for participants and investigators
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- functional yogurt (Experimental): Participants are given the symbiotic yogurt daily (180 ml)
  Interventions: Dietary Supplement: yogurt
- control yogurt (Experimental): Participants are given the control yogurt daily (180 ml)
  Interventions: Dietary Supplement: yogurt

INTERVENTIONS:
Dietary Supplement: yogurt

SUMMARY:
Prebiotics have been linked to increased calcium absorption in animal and human studies (particularly in adolescents and in premenopausal women). Similarly, probiotics have been found to benefit calcium homeostasis in pregnant women, and to promote bio-mineralization in animal models. The effect of symbiotic on calcium absorption has been tested in rats, but not in human studies. The primary objective of this study is to investigate the effect of daily consumption of a functional symbiotic yogurt containing inulin and Lactobacillus rhamnosus compared to a control yogurt, on calcium absorption in young adult women. A secondary objective is to relate changes in calcium absorption following yogurt consumption, with calcium metabolism, vitamin D status, bone mass, calcium intake and overall composition of habitual diet.

DETAILED DESCRIPTION:
A potential strategy to reduce the risk of osteoporosis later in life is to promote optimal bone mass during early adulthood by including in the diet functional foods that maximize the efficiency of calcium absorption. This approach is specially important in women because of their greater risk for osteoporosis than men. In this study, we hypothesized that the daily consumption of a yogurt containing inulin and Lactobacillus rhamnosus (symbiotic yogurt) increases the efficiency of calcium absorption in young adult women when compared to daily consumption of a yogurt of similar composition but without prebiotic or probiotic (control yogurt). Subjects in this study will be randomly assigned to consume daily the symbiotic yogurt or the control yogurt during two 3-week periods with a wash-out period of 3-weeks, in a cross-over design. Calcium absorption will be measured by stable calcium isotope methodology. Bone mass (BMD, BMC) will be measured by dual-Y ray absorptiometry. Serum intact parathyroid hormone, 25-hydroxyvitamin D and dietary intake will be measured by conventional methods.

ELIGIBILITY:
Inclusion Criteria:

* ages 18 to 35 years
* generally healthy

Exclusion Criteria:

* pregnancy/lactation
* BMI <18,5 kg/m2
* BMI> 29 kg/m2
* metabolic disorders, bone, liver or kidney disease that may affect calcium metabolism
* smoking

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in calcium absorption | Day 21 and Day 63
  Fractional calcium absorption measured with stable isotopes

SECONDARY OUTCOMES:
Serum 25(OH) vitamin D | Day 1
  Serum 25 (OH) vitamin D values expressed in nmol/liter
Bone mineral content and bone mineral density | Day 1
  Bone mineral content and bone mineral density values expressed as Z scores.
Dietary calcium intake | Day 1
  Values expressed in mg/d

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cornes R, Sintes C, Pena A, Albin S, O'Brien KO, Abrams SA, Donangelo CM. Daily Intake of a Functional Synbiotic Yogurt Increases Calcium Absorption in Young Adult Women. J Nutr. 2022 Jul 6;152(7):1647-1654. doi: 10.1093/jn/nxac088. PMID 35411924